CLINICAL TRIAL: NCT02164916
Title: Randomized Phase II Study of Irinotecan and Cetuximab With or Without Vemurafenib in BRAF Mutant Metastatic Colorectal Cancer
Brief Title: S1406 Phase II Study of Irinotecan and Cetuximab With or Without Vemurafenib in BRAF Mutant Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S1406; U10CA180888 (NIH); S1406 (Other: SWOG); NCI-2014-00814 (Other: NCI)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer
Keywords: BRAF Mutant; Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Immunoglobulin G; Disulfides; Irinotecan; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cetuximab, irinotecan hydrochloride) (Active Comparator): Patients receive cetuximab IV and irinotecan hydrochloride IV on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross over to Arm II.
  Interventions: Biological: cetuximab; Drug: irinotecan hydrochloride
- Arm II (cetuximab, irinotecan hydrochloride, vemurafenib) (Experimental): Patients receive cetuximab and irinotecan hydrochloride as in Arm I and vemurafenib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: irinotecan hydrochloride; Drug: vemurafenib

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: 11460; 205923-56-4; 3610; 714692; Anti-EGFR Monoclonal Antibody; Anti-Epidermal Growth Factor Receptor Monoclonal Antibody; C225; C225 monoclonal antibody; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225; Immunoglobulin G1; anti-(human epidermal growth factor receptor) (human-mouse monoclonal C225 gamma1-chain); disulfide with human-mouse monoclonal C225 kappa-chain; dimer; MOAB C225; monoclonal antibody C225
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; camptothecin-11; CPT-11; irinotecan; irinotecan HCl; U-101440E
Drug: vemurafenib — Given PO
  Other Names: BRAF(V600E) kinase inhibitor RO5185426; PLX4032; RG7204; RO5185426; Zelboraf
  Arms: Arm II (cetuximab, irinotecan hydrochloride, vemurafenib)

SUMMARY:
This randomized phase II trial studies how well irinotecan hydrochloride and cetuximab with or without vemurafenib works in treating patients with colorectal cancer that has spread to nearby tissue or lymph nodes, that has spread to other places in the body, or cannot be removed by surgery. Irinotecan hydrochloride and vemurafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, may block the ability of tumor cells to grow and spread. It is not yet known whether irinotecan hydrochloride and cetuximab are more effective with or without vemurafenib in treating colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival (PFS) of v-raf murine sarcoma viral oncogene homolog B (BRAF) mutant metastatic colorectal cancer patients treated with irinotecan (irinotecan hydrochloride), cetuximab, and vemurafenib, compared to a control arm of irinotecan and cetuximab.

SECONDARY OBJECTIVES:

I. To evaluate the frequency and severity of toxicity associated with each of the treatment arms in this patient population.

TERTIARY OBJECTIVES:

I. To evaluate overall survival (OS) in treatment Arms 1 and 2. II. To evaluate the overall response rate (ORR), including confirmed and unconfirmed, complete and partial response, in treatment Arms 1 and 2 in the subset of patients with measurable disease.

III. To estimate rates of OS, ORR, and PFS in patients who register to Arm 3 after disease progression on Arm 1.

IV. To evaluate low-frequency Kirsten rat sarcoma viral oncogene homolog (KRAS) or neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS) mutations as detected by high-depth sequencing as predictive biomarkers of efficacy.

V. To evaluate phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) pathway activation through PIK3CA mutations or phosphatase and tensin homolog (PTEN) protein loss as a predictive biomarker of innate resistance to this regimen.

VI. To evaluate gene expression signatures from screened patients with v-raf murine sarcoma viral oncogene homolog B wild type (BRAFWT) and BRAFV600E tumors.

VII. To provide validation of BRAF immunohistochemistry (IHC) using complementary sequencing methodology from screened patients with BRAFWT and BRAFV600E tumors.

VIII. To confirm the estimated sensitivity of detectable BRAF V600E circulating cell-free deoxyribonucleic acid (DNA) as a non-invasive biomarker for BRAF V600E mutation as detected by IHC in the primary tumor.

IX. To correlate radiographic tumor response with change in quantification of BRAFV600E alleles in circulating cell-free DNA.

X. To monitor for known mechanism of acquired resistance to epidermal growth factor receptor (EGFR) inhibition in circulating cell-free DNA (KRAS, NRAS mutations).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cetuximab intravenously (IV) and irinotecan hydrochloride IV on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross over to Arm II.

ARM II: Patients receive cetuximab and irinotecan hydrochloride as in Arm I and vemurafenib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-6 months for 3 years.

ELIGIBILITY:
* STEP I INITIAL REGISTRATION: BRAFV600E TESTING:
* Patients must have histologically or cytologically documented adenocarcinoma of the colon or rectum that is either metastatic, or locally advanced and unresectable
* Patients must have BRAFV600E mutant status documented by a Clinical Laboratory Improvements Amendments (CLIA) certified laboratory on a pathology report prior to Step 2 registration; use of an Food and Drug Administration (FDA)-approved test is preferred although other BRAF tests at a CLIA-certified laboratory may also be accepted; if a BRAFV600E mutation is known, then the patient must be registered to Step 2 Randomization immediately following Step 1 Initial Registration; if testing has not been performed locally, BRAFV600E testing must be completed by the central lab prior to Step 2 Randomization; if the specimen does not have a BRAFV600E mutation, the patient is ineligible for Step 2 Randomization
* Brain metastases are allowed if they have been adequately treated with radiotherapy or surgery and stable for at least 90 days prior to Step 1 Initial Registration; eligible patients should be neurologically asymptomatic and without corticosteroid treatment for at least 7 days prior to Step 1 Initial Registration
* Patients must have had one or two prior regimens of systemic chemotherapy for metastatic disease; prior treatment with irinotecan is allowed; a maintenance regimen of 5-fluorouracil or capecitabine, with or without bevacizumab, should not be counted as a separate line of treatment; prior treatment for metastatic disease is not required for patients who experienced disease recurrence during or within 6 months of completion of adjuvant chemotherapy
* Patients must not have been treated with any of the following prior to Step 2 Randomization:

  * Cetuximab, panitumumab, or any other monoclonal antibody against EGFR or inhibitor of EGFR
  * BRAF inhibitor including, but not limited to, vemurafenib or dabrafenib; regorafenib is not considered a BRAF inhibitor for the purpose of determining trial eligibility
  * Mitogen-activated protein/extracellular signal-regulated kinase (MEK) inhibitor including, but not limited to, trametinib or selumetinib
* Previous chemotherapy, immunotherapy, or radiation therapy must have been completed at least 14 days prior to Step 1 Initial Registration and all toxicity must be resolved to Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) grade 1 (with the exception of CTCAE v4.0 grade 2 neuropathy) prior to Step 1 Initial Registration
* Patients must not have a tumor with a mutation detected in codons 12 or 13 in KRAS; patients must not have a tumor with a known mutation detected in codons 61, 117, or 146 of KRAS or NRAS
* SPECIMEN SUBMISSION CRITERIA:
* Patients must have tumor (slides or block) available for submission for V600E BRAF testing
* Patients must have additional tumor available and be willing to submit tissue and blood samples
* SPECIMEN SUBMISSION CRITERIA REGULATORY CRITERIA:
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines; for Step 1 Initial Registration of patients who have not yet submitted specimens for the central BRAFV600E testing, the appropriate consent form is the Step 1 Consent Form; for both Step 1 Initial Registration and Step 2 Randomization of patients whose BRAF mutation status is already known, the appropriate consent form is the Step 2 Consent Form
* STEP 2 RANDOMIZATION:
* Patients must have BRAFV600E mutation
* Patients must have measurable or non-measurable metastatic disease; computed tomography (CT) scans or magnetic resonance imaging (MRIs) used to assess all disease must have been completed within 28 days prior to Step 2 Randomization; CT scans or MRIs must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Patients must have a Zubrod performance status of 0-1
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,00/mcL
* Hemoglobin >= 9 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (IULN) or =< 5 x IULN if liver metastases are present
* Total bilirubin =< 1.5 x IULN
* Serum creatinine =< 1.5 x IULN within 14 days prior to Step 2 Randomization OR
* Calculated creatinine clearance > 60 ml/min; the serum creatinine value used in the calculation must have been obtained within 14 days prior to Step 2 Randomization
* Patients must have an electrocardiogram (ECG) within 14 days prior to Step 2 Randomization
* Patients must have corrected QT (QTc) =< 500 msec
* Patients must not have a known history of Gilbert's Syndrome or known homozygosity for the UDP glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1)*28 allele
* Patients must not have interstitial pneumonia or extensive symptomatic interstitial fibrosis of the lung
* Patients must not have an uncontrolled intercurrent illness including, but not limited to, active bleeding diathesis, uncontrolled infection/disorders, nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy, or psychiatric illness/social situations which would limit compliance with study requirements
* Patients must be able to swallow pill/tablet and have no refractory nausea, vomiting, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate absorption
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method while on study and for 30 days after study treatment; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures, he/she is responsible for beginning contraceptive measures
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years
* STEP 2 RANDOMIZATION REGULATORY CRITERIA:
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines; for all patients, the appropriate consent form for this registration is the Step 2 Consent Form
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 3 CROSSOVER REGISTRATION:
* Patients must have documented disease progression while on Arm 1 of this protocol; the follow-up tumor assessment form documenting disease progression must be submitted to Southwestern Oncology Group (SWOG) prior to Step 3
* Registration to Step 3 Crossover must be within 28 days of discontinuation of Arm 1 protocol treatment; patients going off treatment for any other reason are not eligible
* ANC >= 1,500/mcL within 14 days prior to Step 3 registration
* Platelets >= 100,00/mcL within 14 days prior to Step 3 registration
* Hemoglobin >= 9 g/dL within 14 days prior to Step 3 registration
* AST and ALT =< 2.5 x institutional upper limit of normal (IULN) or =< 5 x IULN if liver metastases are present within 14 days prior to Step 3 registration
* Total bilirubin =< 1.5 x IULN within 14 days prior to Step 3 registration
* Serum creatinine =< 1.5 x IULN within 14 days prior to Step 3 registration OR
* Calculated creatinine clearance > 60 ml/min; the serum creatinine value used in the calculation must have been obtained within 14 days prior to Step 3 registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11-13 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund S Kopetz, M.D., Principal Investigator — M.D. Anderson
Locations (763):
- United States (763):
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Mercy Cancer Center-Hot Springs, Hot Springs, Arkansas
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - PCR Oncology, Pismo Beach, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Medical Oncology and Hematology Group PC-Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Florida Hospital Cancer Institute Altamonte, Altamonte Springs, Florida
  - University of Florida, Gainesville, Florida
  - Florida Hospital Kissimmee, Kissimmee, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Florida Urology Associates-Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Florida Hospital East Orlando, Orlando, Florida
  - Florida Hospital Cancer Institute Winter Park, Winter Park, Florida
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Leeward, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Porter Memorial Hospital, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Story County Medical Center-South Campus, Nevada, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren-Bay Region, Bay City, Michigan
  - Henry Ford Cancer Institute¿Downriver, Brownstown, Michigan
  - Great Lakes Cancer Institute, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Assarian Cancer Center, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Medical Offices West, Norfolk, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hemotology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Weill Medical College of Cornell University, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Scotland Memorial Hospital-Laurinburg Cancer Center, Laurinburg, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH-Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center, Williamsport, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Scott and White Healthcare Round Rock, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Wheaton Franciscan Healthcare - Saint Joseph, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming

REFERENCES:
- [Derived] Kopetz S, Guthrie KA, Morris VK, Lenz HJ, Magliocco AM, Maru D, Yan Y, Lanman R, Manyam G, Hong DS, Sorokin A, Atreya CE, Diaz LA, Allegra C, Raghav KP, Wang SE, Lieu CH, McDonough SL, Philip PA, Hochster HS. Randomized Trial of Irinotecan and Cetuximab With or Without Vemurafenib in BRAF-Mutant Metastatic Colorectal Cancer (SWOG S1406). J Clin Oncol. 2021 Feb 1;39(4):285-294. doi: 10.1200/JCO.20.01994. Epub 2020 Dec 23. PMID 33356422

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Cetuximab, Irinotecan Hydrochloride) | Arm II (Cetuximab, Irinotecan Hydrochloride, Vemurafenib)
Started | 52 | 54
Eligible | 50 | 49
Cross-over to Arm II | 24 (Following disease progression on Arm 1. Note: these patients are also counted in 'Not Completed'.) | 0
Completed | 0 | 0
Not Completed | 52 | 54
Not completed — Adverse Event | 3 | 8
Not completed — Death | 1 | 1
Not completed — Refusal unrelated to adverse event | 3 | 7
Not completed — Progression | 37 | 26
Not completed — Not protocol specified | 5 | 1
Not completed — Reason under review | 1 | 6
Not completed — Not eligible | 2 | 5

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cetuximab, Irinotecan Hydrochloride) | Arm II (Cetuximab, Irinotecan Hydrochloride, Vemurafenib) | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Median (Full Range); unit: years] | 62 [31 to 83] | 60 [34 to 83] | 62 [31 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 21 | 58
  Male | 13 | 28 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 48 | 46 | 94
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 49 | 43 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Prior treatment with Irinotecan [Number; unit: participants]
  Yes | 19 | 20 | 39
  No | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: From date of randomization to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact. Progression is defined as one or more of the following: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm; unequivocal progression of non-measurable disease in the opinion of the treating physician; appearance of any new lesion/site; and/or death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Up to 3 years from randomization
Population: Eligible and analyzable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cetuximab, Irinotecan Hydrochloride) | Arm II (Cetuximab, Irinotecan Hydrochloride, Vemurafenib)
Number analyzed (Participants) | 50 | 49
months | 2.0 [1.8 to 2.1] | 4.3 [3.6 to 5.7]
Statistical Analysis 1: Comparison: Arm I (Cetuximab, Irinotecan Hydrochloride) vs Arm II (Cetuximab, Irinotecan Hydrochloride, Vemurafenib); Test type: Superiority; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.31 to 0.75]

2. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary.
Measure: Number; unit: Participants
Groups:
- Cetuximab + Irinotecan: Patients receive cetuximab IV and irinotecan hydrochloride IV on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Vemurafenib + Cetuximab + Irinotecan; Crossover: Vemurafenib + Cetuximab + Irinotecan: Patients receive cetuximab IV and irinotecan hydrochloride IV on days 1 and 14, and vemurafenib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Cetuximab + Irinotecan | Vemurafenib + Cetuximab + Irinotecan | Crossover: Vemurafenib + Cetuximab + Irinotecan
Number analyzed (Participants) | 46 | 46 | 21
Participants
  Abdominal pain | 1 | 2 | 0
  Alkaline phosphatase increased | 2 | 0 | 1
  Allergic reaction | 1 | 0 | 0
  Anaphylaxis | 1 | 0 | 0
  Anemia | 0 | 6 | 1
  Anorexia | 2 | 3 | 0
  Arthralgia | 0 | 3 | 0
  Arthritis | 0 | 0 | 1
  Blood bilirubin increased | 1 | 0 | 1
  Cardiac disorders - Other, specify | 0 | 0 | 1
  Colitis | 0 | 0 | 1
  Colonic obstruction | 1 | 0 | 0
  Creatinine increased | 0 | 1 | 0
  Dehydration | 3 | 5 | 0
  Diarrhea | 6 | 11 | 7
  Electrocardiogram QT corrected interval prolonged | 0 | 1 | 1
  Fatigue | 7 | 7 | 7
  Febrile neutropenia | 2 | 5 | 0
  Gastric hemorrhage | 0 | 0 | 1
  Generalized muscle weakness | 1 | 1 | 1
  Hyperkalemia | 0 | 0 | 1
  Hypocalcemia | 0 | 0 | 1
  Hypokalemia | 1 | 5 | 2
  Hypomagnesemia | 2 | 0 | 1
  Hyponatremia | 1 | 2 | 0
  Infusion related reaction | 1 | 1 | 0
  Insomnia | 0 | 0 | 1
  Lower gastrointestinal hemorrhage | 0 | 0 | 1
  Lung infection | 0 | 1 | 0
  Lymphocyte count decreased | 0 | 1 | 0
  Metabolic acidosis | 1 | 0 | 0
  Mucositis oral | 0 | 2 | 0
  Myalgia | 0 | 2 | 0
  Nausea | 1 | 9 | 1
  Neutrophil count decreased | 3 | 15 | 2
  Pain | 0 | 1 | 0
  Palmar-plantar erythrodysesthesia syndrome | 0 | 0 | 1
  Pancreatitis | 0 | 1 | 0
  Papulopustular rash | 1 | 0 | 0
  Photosensitivity | 0 | 1 | 0
  Platelet count decreased | 0 | 1 | 0
  Pruritus | 1 | 0 | 0
  Rash acneiform | 3 | 0 | 0
  Rash maculo-papular | 0 | 1 | 1
  Rash pustular | 0 | 1 | 0
  Sepsis | 0 | 2 | 0
  Thromboembolic event | 0 | 0 | 1
  Treatment related secondary malignancy | 0 | 0 | 1
  Urinary tract infection | 1 | 0 | 1
  Vomiting | 1 | 5 | 0
  Weight loss | 1 | 0 | 0
  White blood cell decreased | 0 | 8 | 2

3. Other Pre Specified Outcome: Overall Survival
Description: From date of randomization to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 3 years from randomization
Population: Eligible and analyzable patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cetuximab, Irinotecan Hydrochloride) | Arm II (Cetuximab, Irinotecan Hydrochloride, Vemurafenib)
Number analyzed (Participants) | 50 | 49
months | 5.9 [3.0 to 9.9] | 9.6 [7.5 to 13.1]

4. Other Pre Specified Outcome: Overall Response Rate
Description: Confirmed response (CR) is two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Partial response (PR) is two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration. Unconfirmed CR is one objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 3 years from randomization
Population: All eligible and analyzable patients with measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cetuximab, Irinotecan Hydrochloride) | Arm II (Cetuximab, Irinotecan Hydrochloride, Vemurafenib)
Number analyzed (Participants) | 47 | 44
Participants
  Partial Response | 1 | 3
  Unconfirmed Partial Response | 1 | 4
  Stable/No Response | 8 | 22
  Increasing Disease | 25 | 7
  Symptomatic Deterioration | 6 | 1
  Assessment Inadequate | 6 | 7

5. Other Pre Specified Outcome: Progression-free Survival in Patients Who Register to Arm 3 (Crossover) After Disease Progression on Arm 1
Description: From date of Step 3 Crossover registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive without report of progression are censored at date of last contact. Progression is defined as one or more of the following: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm; unequivocal progression of non-measurable disease in the opinion of the treating physician; appearance of any new lesion/site; and/or death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Up to 3 years from randomization
Population: All eligible and analyzable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crossover: Vemurafenib + Cetuximab + Irinotecan
Number analyzed (Participants) | 22
months | 5.8 [2.8 to 6.1]

6. Other Pre Specified Outcome: Overall Survival in Patients Who Register to Arm 3 (Crossover) After Disease Progression on Arm 1
Description: as for outcome 3
Time Frame: Up to 3 years from randomization
Population: Eligible and analyzable patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crossover: Vemurafenib + Cetuximab + Irinotecan
Number analyzed (Participants) | 22
months | 12.1 [4.5 to 12.5]

7. Other Pre Specified Outcome: Overall Response Rate in Patients Who Register to Arm 3 (Crossover) After Disease Progression on Arm 1
Description: as for outcome 4
Time Frame: Up to 3 years from randomization
Population: Eligible and analyzable patients with measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover: Vemurafenib + Cetuximab + Irinotecan
Number analyzed (Participants) | 18
Participants
  Partial Response | 2
  Unconfirmed Partial Response | 1
  Stable/No Response | 10
  Increasing Disease | 5

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Eligible patients who received any treatment and were assessed for adverse events are included in the adverse event summaries.
Arm/Group | Cetuximab + Irinotecan | Vemurafenib + Cetuximab + Irinotecan | Crossover: Vemurafenib + Cetuximab + Irinotecan
All-Cause Mortality (participants affected / at risk) | 3/46 | 4/46 | 2/21
Serious Adverse Events (participants affected / at risk) | 3/46 | 25/46 | 10/21
Other Adverse Events (participants affected / at risk) | 45/46 | 41/46 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Irinotecan (N=46) | Vemurafenib + Cetuximab + Irinotecan (N=46) | Crossover: Vemurafenib + Cetuximab + Irinotecan (N=21)
Anemia (Blood and lymphatic system disorders) | 0 | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac disorders-Other (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 5 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Jejunal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 5 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 5 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1
Death NOS (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 1
Fever (General disorders) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 4 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2
Alkaline phosphatase increased (Investigations) | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 1 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 3 | 0
White blood cell decreased (Investigations) | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 5 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Irinotecan (N=46) | Vemurafenib + Cetuximab + Irinotecan (N=46) | Crossover: Vemurafenib + Cetuximab + Irinotecan (N=21)
Anemia (Blood and lymphatic system disorders) | 11 | 21 | 9
Blurred vision (Eye disorders) | 1 | 4 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 2
Eye disorders-Other (Eye disorders) | 1 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 19 | 18 | 5
Colonic obstruction (Gastrointestinal disorders) | 3 | 0 | 1
Constipation (Gastrointestinal disorders) | 11 | 3 | 4
Diarrhea (Gastrointestinal disorders) | 27 | 28 | 16
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1
Hemorrhoids (Gastrointestinal disorders) | 3 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 7 | 19 | 5
Nausea (Gastrointestinal disorders) | 27 | 27 | 16
Vomiting (Gastrointestinal disorders) | 14 | 21 | 6
Edema limbs (General disorders) | 3 | 8 | 4
Fatigue (General disorders) | 31 | 32 | 16
Fever (General disorders) | 2 | 9 | 2
Infusion related reaction (General disorders) | 4 | 3 | 1
Pain (General disorders) | 3 | 4 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1
Alanine aminotransferase increased (Investigations) | 10 | 3 | 4
Alkaline phosphatase increased (Investigations) | 11 | 7 | 7
Aspartate aminotransferase increased (Investigations) | 12 | 4 | 5
Blood bilirubin increased (Investigations) | 3 | 7 | 2
Creatinine increased (Investigations) | 1 | 4 | 0
INR increased (Investigations) | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 4 | 3
Neutrophil count decreased (Investigations) | 11 | 20 | 8
Platelet count decreased (Investigations) | 5 | 3 | 0
Weight loss (Investigations) | 6 | 13 | 3
White blood cell decreased (Investigations) | 8 | 15 | 5
Anorexia (Metabolism and nutrition disorders) | 13 | 14 | 5
Dehydration (Metabolism and nutrition disorders) | 10 | 2 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 5 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 8 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 12 | 20 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 20 | 12 | 11
Hyponatremia (Metabolism and nutrition disorders) | 5 | 10 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 14 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 7 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 9 | 2
Dizziness (Nervous system disorders) | 4 | 6 | 2
Dysgeusia (Nervous system disorders) | 2 | 4 | 2
Headache (Nervous system disorders) | 5 | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 9 | 3
Anxiety (Psychiatric disorders) | 2 | 3 | 1
Depression (Psychiatric disorders) | 1 | 5 | 0
Insomnia (Psychiatric disorders) | 5 | 4 | 2
Hematuria (Renal and urinary disorders) | 2 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 15 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 8 | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 3 | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 11 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 27 | 22 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 13 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 8 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hot flashes (Vascular disorders) | 0 | 3 | 1
Hypertension (Vascular disorders) | 4 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT02164916/Prot_SAP_ICF_000.pdf